CLINICAL TRIAL: NCT06811545
Title: Exploring the Effects of Multi-Joint Neuromuscular Electrical Stimulation on Training Gait of Children With Cerebral Palsy
Brief Title: Evaluating the Effects of an Electrical Stimulator on Improving the Walking Ability of Children With Cerebral Palsy
Acronym: CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0406-24-FB; P20GM109090 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy Children; Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Cerebral Palsy Group (Experimental): The Cerebral Palsy Group (CP), intervention group, will receive a low power electrical stimulation, Neuromuscular Electrical Stimulation (NMES), on different combination of their lower limb muscles while walking on the treadmill.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES)
- Healthy Adults Group (Active Comparator): The Healthy Adults Group (HA) will receive a similar low power electrical stimulation, Neuromuscular Electrical Stimulation (NMES), as that received by the Cerebral Palsy Group. However, they will will only receive NMES in specific muscle groups and the only variable across conditions will be the power of stimulation.
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES)

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (NMES) — Children with CP can have trouble with daily tasks such as walking. This raises their risk of disability as they age into their teens. Current treatments are not very effective. In this study, children with CP will walk on a treadmill while receiving NMES on their lower limb muscles, using surface electrodes, while their gait dynamics are assessed. Our proposed study aims to gather preliminary evidence to support the potential efficacy of NMES assistance to muscles across all lower limb joints during walking, i.e., multi-joint NMES assistance. Additionally, the investigators aim to investigate the optimal level of intensity.

SUMMARY:
The goal of this study is to see if gentle electrical stimulation can help children with cerebral palsy (CP) walk more easily. This stimulation, called neuromuscular electrical stimulation (NMES), sends small pulses to muscles to help them activate. Researchers will test different ways of using NMES to find out which method works best.

Participants will walk on a treadmill at a comfortable speed while NMES is applied to leg muscles. The study will compare different stimulation settings to see which one helps the most.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) can have trouble with daily tasks such as walking. This raises their risk of disability as they age into their teens. Current treatments are not very effective. In this study, children with CP will walk on a treadmill while receiving neuromuscular electrical stimulation (NMES) on their lower limb muscles, using surface electrodes, while gait dynamics are assessed. The proposed study aims to gather preliminary evidence to support the potential efficacy of NMES assistance to muscles across all lower limb joints during walking, i.e., multi-joint NMES assistance. Additionally, the study aims to investigate the optimal level of intensity. Investigators intend to quantify neuroprosthetic, i.e., immediate effects during NMES assistance on gait kinematics.

Up to 36 children between the ages of 7 to 18 who are diagnosed with spastic diplegic cerebral palsy and GMFCS level 1 - 3 will be recruited for this study. The study consists of two assessment sessions. During all sessions, the participants will walk on a treadmill with and without NMES assistance at self selected walking speed. The assessment sessions consist of multiple NMES conditions. Each condition lasts about 1 minute and will be repeated 3 times, with 30 seconds rest between trials for each condition and 5 minutes between each condition. The total walking time will not exceed 30 minutes. Each visit will last about 3 hours. The assessment sessions will begin with a no-stimulation condition and follow with multiple NMES conditions consisting of NMES assistance to various lower limb muscle combinations.

With the aim of developing our NMES system and improving result feasibility, we will recruit up to 15 healthy adults aged between 20 and 40 before involving CP subjects. They will undergo a similar procedure as the CP group with a maximum of 2 sessions. However, unlike the CP group, they will not be exposed to multiple NMES conditions. Instead, they will receive NMES only on a specific muscle combination. The only difference across the conditions will be the intensity of the stimulation: participants will experience either no stimulation, sensory-level stimulation, or motor threshold (MT) stimulation.

ELIGIBILITY:
*Inclusion Criteria*

CP Group:

* Age 7-18
* Diagnosis of spastic diplegic cerebral palsy (CP)
* GMFCS level I-III (be able to walk with or without assistive devices)
* MIGR < 40% femoral head covering in acetabulum
* Crouch, equinus, or jump gait
* At least 0° passive dorsiflexion range of motion (ROM)
* Sufficient visuoperceptual, cognitive, and communication skills
* Seizure-free or well-controlled seizures
* No other neurological or musculoskeletal disorders (e.g. dystonia, severe scoliosis, hip instability
* Ability to travel to the University of Nebraska at Omaha two times
* Ability to communicate pain or discomfort
* Ability to obtain child assent and obtain parent/guardian consent

Healthy adults (control) group:

* Adults aged 20 to 40
* Adults with good physical health
* Adults with the ability to follow verbal instructions
* Adults with the ability to walk on a treadmill for 15 minutes
* No orthopedic surgery on the lower limb within the past 3 months

*Exclusion Criteria*

CP Group:

* Diagnosis of athetoid or ataxic cerebral palsy (CP)
* Scoliosis with primary curve > 49%
* Spinal fusions extending into the pelvis
* Lower Extremity (LE) joint instability or dislocation
* Severe tactile hypersensitivity
* LE botulinum injections in the past 6 mo
* Implanted medical device contraindicative of functional electrical stimulation (FES)
* Pregnancy
* Severe LE spasticity (Modified Ashworth Scale score of 4 or greater)
* History of pulmonary disease limiting exercise tolerance (Asthma Control Test screen)
* History of cardiac disease (American Heart Association, AH,) screen)
* Excessive LE joint pain during walking
* Severely limited range of joint motion/ irreversible muscle contractures, i.e.> 10° knee flexion, >15° hip flexion contractures, or >5° plantarflexion contractures
* LE surgery or significant injury within 1 yr.

Healthy adults (control) group:

* Adults with any chronic illnesses or medical conditions that could impact their health.
* Adults with significant behavioral or emotional issues that could indicate developmental disorders or psychological conditions.
* Adults with diagnosed developmental disorders (e.g., autism, ADHD, learning disabilities)
* Adults with surgery on their lower limb within the past 3 months.

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Gait Variable Index (GDI) | Baseline (enrollment) and the end of assessment at 3 weeks
  Gait Variable Index (GDI) is an index of gait pathology based on 15 different kinematic measures (bilaterally) or nine unilaterally. The GDI score ranges from 0 to 100 where 100 represents atypically developing's (TD) normal GDI score.

CONTACTS AND LOCATIONS:
Overall Officials: Ahad Behboodi, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Biomechanics Research Building, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No